CLINICAL TRIAL: NCT05549570
Title: Single Dose Crossover Comparative Bioavailability Study of Metformin/Sitagliptin 850 mg/50 mg Film-coated Tablets in Healthy Male and Female Volunteers.
Brief Title: Comparative Bioavailability Study of Metformin/Sitagliptin 850 mg/50 mg Tablets in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galenicum Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GLU-P6-810
Record Dates: First submitted 2022-09-16; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Bioequivalence; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference group (Experimental): Thirty minutes after the start of the breakfast, a single dose of the Reference formulation was administered with approximately 240 mL of water at ambient temperature
  Interventions: Drug: Sitagliptin/Metformin HCl 50/850 mg film-coated tablet
- Test group (Experimental): Thirty minutes after the start of the breakfast, a single dose of the Test formulation was administered with approximately 240 mL of water at ambient temperature
  Interventions: Drug: Sitagliptin/Metformin HCl 50/850 mg film-coated tablet

INTERVENTIONS:
Drug: Sitagliptin/Metformin HCl 50/850 mg film-coated tablet — The subjects randomly received single oral dose of Sitagliptin/Metformin HCl 50/850 mg film-coated tablet

SUMMARY:
The objective of this study was to evaluate and compare the bioavailability and therefore to assess the bioequivalence of two different formulations of metformin/sitagliptin after a single oral dose administration under fed conditions.

ELIGIBILITY:
The main Inclusion Criteria were:

* non- or ex-smokers
* body mass index (BMI) within 18.5 to 30.0 kg/m2, inclusively
* no clinically significant abnormality found in the 12-lead electrocardiogram (ECG) performed at study entry
* negative pregnancy test for female subjects
* healthy according to medical history, complete physical examination (including vital signs) and laboratory tests (general biochemistry, hematology and urinalysis)

Exclusion Criteria:

* Females who were pregnant or were lactating
* History of significant hypersensitivity to metformin, sitagliptin or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease that may have affected drug bioavailability
* Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
* History of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
* Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >119 msec and QTc > 450 msec for males and QTc > 460 for females) on the screening ECG or other clinically significant ECG abnormalities
* Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study
* Any history of tuberculosis and/or prophylaxis for tuberculosis
* Positive screening of alcohol and/or drugs of abuse
* Positive results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or Hepatitis C Virus (HCV (C)) tests
* Females who were pregnant according to a positive pregnancy test
* Volunteers who took metformin and/or sitagliptin in the previous 28 days before day 1 of this study
* Volunteers who took an Investigational Product (in another clinical trial) in the previous 28 days before day 1 of this study
* Volunteers who had already participated in this clinical study
* Volunteers who donated 50 mL or more of blood in the previous 28 days before day 1 of this study
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-22 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 48 hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) 0-t | 48 hours
  Evaluation of plasma concentration-time curve from zero to the time of the last measurable time point t

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs), abnormal clinical laboratory test results, physical examination findings and glycemia. | 1 week
  Adverse events were classified by System Organ Class (SOC) and Preferred Term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA), version 20.1 (Medrio database) and graded as mild, moderate, or severe.
  The principal investigator or qualified designee determined the relationship of any AE to the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schnaars Y, Gaikwad S, Gottwald-Hostalek U, Uhl W, Ribot O, Varanasi KVS, Rodriguez L, Torrejon J, Gomez L. Bioequivalence Evaluation in Healthy Volunteers: New Generic Formulations of Sitagliptin and Sitagliptin-Metformin Fixed-Dose Combination Compared with the Originator Products. Diabetes Ther. 2023 Feb;14(2):347-362. doi: 10.1007/s13300-022-01349-2. Epub 2022 Dec 16. PMID 36526947